CLINICAL TRIAL: NCT07366879
Title: Randomised Controlled Trial of Exercise Intervention as an Adjunct to Medical Therapy in Newly Diagnosed Patients With Pulmonary Arterial Hypertension
Brief Title: Exercise Intervention as an Adjunct to Medical Therapy in Newly Diagnosed Patients With Pulmonary Arterial Hypertension
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Golden Jubilee National Hospital (Other Government)
Collaborators: Chiesi Farmaceutici S.p.A. (Industry); University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 25/CARD/29
Record Dates: First submitted 2026-01-07; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: pulmonary arterial hypertension; PAH; pulmonary hypertension; exercise training; exercise adherence
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary

STUDY DESIGN:
Intervention Model Description: More fitting to a Waitlist Randomised Control Trial as participants are assigned to an intervention or control group initially, but the control group will go on to receive the intervention at a later time, whereas the intervention group will be allowed to continue exercising. Therefore not strictly a crossover trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Exercise Intervention Group then Adherence package group during follow-up phase (Experimental): Initially randomised to the exercise intervention group. Following completion of the exercise intervention, then randomised to receive the adherence support package.
  Interventions: Other: Home-based, remotely delivered, supervised Exercise programme
- Exercise Intervention Group then control group during follow-up phase (Experimental): Initially randomised to the exercise intervention group. Following completion of the exercise intervention, then randomised to the control group during the follow-up phase, so not given the adherence support package.
  Interventions: Other: Home-based, remotely delivered, supervised Exercise programme
- Control group, then the Adherence package group during the follow-up phase (No Intervention): Initially randomised to the control group. Then randomised to receive the adherence support package in the follow-up phase
- Control group, then also randomised to the control group in the follow-up phase (No Intervention): Initially randomised to the control group. Following completion of the exercise intervention, then randomised to be in the control group in follow-up phase, so not given the adherence support package.

INTERVENTIONS:
Other: Home-based, remotely delivered, supervised Exercise programme — A home-based remotely delivered supervised exercise programme
  Arms: Exercise Intervention Group then Adherence package group during follow-up phase; Exercise Intervention Group then control group during follow-up phase

SUMMARY:
The goal of this clinical trial is to learn if an exercise programme started shortly after diagnosis improves the fitness and mental wellbeing of patients with pulmonary hypertenion over and above medication alone. It will also learn about whether extra support can help patients keep up with exercise in the long term. The main questions it aims to answer are:

* Doe exercise improve how far patients can walk over six minutes
* Does exercise improve quality of life scores
* Does exercise improve mental health scores
* Does extra support after an exercise programme help patients to continue exercising in the long term

Researchers will compare the exercise programme to a control group (a group of similar patients who do not receive the exercise programme) to see the effect that exercise has.

Participants in the exercise programme group will:

* Undergo an exercise programme for 12 weeks, starting around 3 months after their diagnosis
* They will undertake the exercise programme at home, remotely supervised by the research team with regular contact
* Visit the clinic at the end of the programme for checkups and tests
* Keep a diary of their exercise and how they are feeling

Participants in the control group will:

-Still undergo the exercise programme, but this will happen at a delayed time, starting around 6 months after diagnosis, to allow for a comparison between the two groups.

Following completion of the exerise programme:

* Half of participants will receive extra support to help them continue to exercise
* The other half will not receive any additional support
* All patients will be reviewed 1 year following the completion of their exercise programme to monitor their ongoing exercise levels.

DETAILED DESCRIPTION:
This study is designed to deliver a remotely supervised, home-based exercise programme to patients newly diagnosed with pulmonary arterial hypertension with a view to early optimisation of their condition. The design is a waitlist randomised controlled trial whereby participants will be randomised to an exercise intervention or control group, with the control group then going on to have access to the exercise programme after a 12-week delay. There will be further randomisation after completion of the exercise programme to determine if participants have access to support package aimed at improving adherence to exercise.

The study objectives are to evaluate:

* The incremental effect of an exercise programme on exercise capacity, quality of life and mental health
* The impact of an additional support package following completion of the exercise programme on adherence to exercise in the long term.

Methodology Patients will be recruited from the Scottish Pulmonary Vascular Unit and consented for the study at the time of diagnosis with pulmonary arterial hypertension.

Participants will be commenced on pulmonary vasodilator therapy as per standard of care decided by the clinical team, then will be reviewed 3 months later at outpatient clinic.

Half of participants will then be randomly assigned to an intervention group and the remaining half to a control group. The intervention group will start a 12-week home-based remotely supervised exercise programme while the control group continue on medical therapy alone to allow for comparison. After this 12 weeks, participants in both groups will be seen back in clinic for further review and data collection. The control group will then commence the exercise programme.

After each participant completes the exercise programme they will then be randomly assigned to either receive a support package from the research team, designed to improve adherence to exercise, or to act as a control group and continue with self-directed exercise. All participants will be reviewed one year after completing the exercise programme to review their adherence to exercise.

Data collection:

Data will be collected at standard of care outpatient clinic appointments (six-minute walk test results, EmPHasis-10 questionnaires, NT-proBNP test. Study questionnaires will also be checked at these visits (PHQ-9 and GAD-7 questionnaires at all visits, exercise adherence rating scale questionnaire at the final visits).

Smartwatches will also be worn by study participants and data will be collected on step count, exercise frequency and intensity, heart rate variability, sleep.

Qualitative data will be gathered from the participants by interview at the end of the exercise programme and following their follow-up phase to evaluate factors that helped or hindered exercise.

Exercise programme:

The exercise programme is carried out fully remotely and has been adopted from the PHAHB study by McCormack et al 2019 and includes induction training sessions (discussing the introduction to exercise equipment, the provided materials, exercise safety and demonstrations) and health coaching sessions (discussing various topics including benefits of exercise, goal setting, action planning, self-monitoring, identification and management of barriers to exercise, problem solving and feedback on behaviour).

There are three types of training activities in the programme which are aerobic training (either walking, cycling or a combination), resistance training (using body weight exercises, but may progress to using resistance bands or light weights) and respiratory training. These activities are built up gradually throughout the programme on an individualised basis over a 12-week period.

Exercise support package:

The exercise adherence package will consist of access to online exercise resources, monthly phone calls from the research team and a forum to allow participant discussion and encouragement.

Sample size: Recruitment target is 40 patients with a 1:1 randomisation to the intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-years-old and above
* Diagnosed with pulmonary hypertension (group I and non-operable group IV) by right heart catheterisation showing:

  * a baseline mean pulmonary artery pressure >20mmHg
  * pulmonary vascular resistance >2 Wood Units
  * pulmonary capillary wedge pressure <15mmHg
* Able to provide written informed consent

Exclusion Criteria:

* Diagnosis with pulmonary hypertension of any other cause

  * Group II (PH due to left heart disease)
  * Group III (PH due to hypoxic lung disease)
  * Operable group IV (PH due to chronic thromboembolic disease amenable to surgical treatment)
  * Group V (unclear and/or multifactorial elements).
* Planned treatment with a research trial medication during the study timeframe
* Consenting clinician and/or patient concern regarding the patient's safety in performing a home-based exercise programme
* Patients with syncopal episodes felt to be related to pulmonary hypertension at time of exercise intervention initiation.
* Severe concurrent medical condition that would prevent participation in study procedures
* Life expectancy <3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-19 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Six-minute walk distance | Around 6 months post diagnosis. (After completion of the exercise programme for those in the intervention group, and on medical therapy alone for those in the control group).
  Distance walked as measured during a six-minute walk test. Measured at around 6 months post-diagnosis to compare those from the exercise intervention group who have just completed their exercise programme, with the control group who have not yet had their exercise programme.

SECONDARY OUTCOMES:
EmPHasis-10 questionnaire | Around 6 months post diagnosis. (After completion of the exercise programme for those in the intervention group, and on medical therapy alone for those in the control group).
  EmPHasis-10 quality of life questionnaire. Minimum value 0, Maximum value 50. Higher scores mean a worse outcome.
NT-proBNP blood test | Around 6 months post diagnosis. (After completion of the exercise programme for those in the intervention group, and on medical therapy alone for those in the control group).
  NTproBNP blood test which is a marker of cardiac strain
Patient Health Questionnaire-9 | Around 6 months post diagnosis. (After completion of the exercise programme for those in the intervention group, and on medical therapy alone for those in the control group).
  Questionnaire validated for evaluating depression- completed by patients. Minimum value 0, Maximum value 27. Higher values indicated a worse outcome.
Generalised Anxiety Disorder 7-item Scale | Around 6 months post diagnosis. (After completion of the exercise programme for those in the intervention group, and on medical therapy alone for those in the control group).
  Questionnaire validated for evaluating anxiety in patients- completed by patients. Minumum value 0, Maximum value 21. Higher scores indicate a worse outcome.

OTHER OUTCOMES:
Exercise adherence rating scale | This will be collected after patients complete the exercise programme and again at the end of their follow-up phase. For patients randomised to Study Group 1, this is at week 37 and week 89 from enrolment. For Study group 2, this is week 25 and week 77.
  Questionnaire validated for evaluating adherence to exercise in patients. Completed by patients. Minimum score 0, Maximum score 24. A higher score indicates better adherence.
Heart rate variability | This will be recorded during recorded sessions by the participant throughout study completion which is on average 83 weeks.
  Variation in time between consecutive heart beats, collected by a smartwatch. Measured in milliseconds. Higher heart rate variability means better fitness and recovery.
Exercise Frequency | This will be recorded during recorded sessions by the participant throughout study completion which is on average 83 weeks.
  Average number of recorded exercise sessions per week, measured as an absolute number. Higher number means more regular exercise.
Exercise Intensity | This will be recorded during recorded sessions by the participant throughout study completion which is on average 83 weeks.
  Exercise intensity is recorded by the participant using a smartwatch during recorded exercise sessions. Exercise intensity is measured by the heart rate during exercise expressed as a percentage of the estimated maximum heart rate. The measure will be recorded as time spent in particular heart rate zones, expressed in hours and minutes. Zone 1: 50-60% of maximum heart rate. Zone 2: 60-70% of maximum heart rate. Zone 3: 70-80% of maximum heart rate. Zone 4: 80-90% of maximum heart rate. Zone 5: 90-100% of maximum heart rate. Longer time spent in higher heart rate zones means higher intensity exercise.
Sleep score | This will be recorded throughout study completion which is on average 83 weeks.
  Sleep score is measured by the smartwatch during sleep and expressed as an absolute value between 0-100. This is calculated based on sleep duration, stages (light, deep or rapid eye movement sleep), movement, and heart rate variability. Higher score means better rest.
Step Count | This will be recorded throughout study completion which is on average 83 weeks.
  Number of steps walked by the participant each day, recorded by the smartwatch. Measured as an absolute value. Higher step count indicates higher activity levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Golden Jubilee National Hospital, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCormack C, Kehoe B, Cullivan S, McCaffrey N, Gaine S, McCullagh B, McCarren A, Hardcastle SJ, Moyna NM. Safety, feasibility and effectiveness of the remotely delivered Pulmonary Hypertension and Home-Based (PHAHB) physical activity intervention. ERJ Open Res. 2024 Jan 8;10(1):00608-2023. doi: 10.1183/23120541.00608-2023. eCollection 2024 Jan. PMID 38264149